CLINICAL TRIAL: NCT06412549
Title: IMPACTO MR: Effect of a Bundle of Interventions on Patients With Central Nervous System Devices - Project Platform Supporting the National Action Plan for Prevention and Control of Antimicrobial Resistance
Brief Title: Effect of a Bundle of Interventions on the Outcomes of Patients With Intracranial Devices (ICP Monitor e EVD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beneficência Portuguesa de São Paulo (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Viviane Cordeiro Veiga, MD, PhD, Principal Investigator, Beneficência Portuguesa de São Paulo
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 6. NUP25000.1672362023-51
Record Dates: First submitted 2024-04-16; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Central Nervous System Infections
Keywords: Bacterial resistance; Health care; Central nervous systen infection; Multi-resistant microorganism
MeSH Terms: conditions — Central Nervous System Infections

STUDY DESIGN:
Intervention Model Description: The first phase of the project included 554 participants (baseline sample) and the second phase included 746 participants (intervention sample). Totaling 1,300 patients with external ventricular drain and/or intracranial pressure monitoring catheter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): Participants over 18 years of age admitted to the ICU in the selected hospitals during the study period, using intracranial pressure monitoring catheters and/or external ventricular drain. Baseline database obtained from the study "Device-related Central Nervous System Infections in Adult Intensive Care Units in Brazil (IMPACTO-SNC)", Carried out during the period from 2022 to 2023.
- Intervention (Experimental): Participants over 18 years old admitted to the ICU in the selected hospitals and trained in the intervention bundle during the study period, using intracranial pressure monitoring catheters and/or external ventricular shunt. Participants included in the period from 2024 to 2026
  Interventions: Behavioral: Health care practices and routines

INTERVENTIONS:
Behavioral: Health care practices and routines — The scope of the project includes a diagnostic visit to participating hospitals, conducted by the coordinating center team, to understand existing protocols related to the management of invasive central nervous system devices (such as intracranial pressure monitoring catheters or external ventricular drains), as well as the physical infrastructure, human resources, and other precautions taken for the prevention and treatment of central nervous system infections. All recommendations in the intervention bundle for patient care will align with the guidelines of the National Health Surveillance Agency (ANVISA) and the best available scientific evidence for preventing infections associated with central nervous system devices.
  * Provide the best care for patients with ICP and/or EVD, based on the best available evidence, with regard to the insertion and maintenance of catheters, as well as diagnosis and treatment in the presence of infection.
  * Training of the multidisciplinary team.
  Arms: Intervention

SUMMARY:
Non-randomized clinical trial conducted in the adult ICUs of Brazilian hospitals participating in the IMPACTO MR Platform, involving adult patients using an intracranial pressure monitoring catheter device or external ventricular drain.

The study will test the hypothesis that the intervention bundle, following ANVISA recommendations for care practices, will reduce the rates of central nervous system infections associated with ICP and EVD devices.

This reduction is expected to lead to more accurate diagnoses, decreased antibiotic usage, shortened ICU and hospital stays, and reduced hospital costs.

DETAILED DESCRIPTION:
IMPACTO MR is a research platform that originated as a prospective and collaborative observational study collecting clinical, microbiological, and cost data from patients admitted to Brazilian adult ICUs during the three-year periods 2018-2020 and 2021-2023. Data were collected from all adult patients admitted to the ICUs of at least 61 hospitals selected for the platform. This project aims to collect data from approximately 20 participating hospitals that perform neurosurgical procedures involving external ventricular drain catheter implantation and intracranial pressure monitoring, with the goal of establishing national data on the prevalence of these conditions.

The first phase of the study will involve completing data collection for the prospective cohort conducted between 2022 and 2023. This cohort is part of the IMPACTO MR: Device-related central nervous system infections in adult intensive care units in Brazil - Action Plan Support Project Platform National Prevention and Control of Antimicrobial Resistance) with the same hospitals. This will represent the baseline incidence of central nervous system infections related to devices and care practices for patients with intracranial pressure monitoring catheters and external ventricular drains. The data will include information on risk factors, care processes, and clinical management in suspected central nervous system infections related to these devices.

In the second phase of the study, an intervention bundle will be implemented to prevent infections and improve care processes in these ICUs progressively. Diagnostic site visits will be conducted at hospitals to support the construction of this intervention bundle, and all participating hospitals will receive continuous training to facilitate measurement of results.

The intervention bundle will be based on ANVISA recommendations for controlling healthcare-associated infections. Currently, the recommendations are based on the care to be followed from pre-operative to post-operative stages, including the use of checklists with daily goals, recommendations for dressing care, catheter handling, and treatment in the presence of infection.

The intervention bundle will be developed by a minimum team of doctors and nurses from the coordinating hospital. After conducting a situational diagnosis, this team will develop care protocols, checklists with daily goals, and training materials for the participating centers.

Throughout the project, systematic feedback meetings will be held to monitor action plans, both remotely and, if necessary, in person.

The intervention will be implemented within each hospital until the proposed sample size is attained.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with intracranial pressure monitoring catheters (intraventricular or intraparenchymal) and/or external ventricular drain.
* The patient can be included from the moment the catheter is implanted, without there being a minimum time for inclusion.

Exclusion Criteria:

* Suspected or confirmed brain death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of the intervention bundle in ICUs on reducing central nervous system infections related to devices. | 30 days after study inclusion
  To compare the incidence of device-related central nervous system infections at baseline and after the implementation of the intervention bundle. The percentage of suspected infection cases and those confirmed by ANVISA criteria will be compared at both study timepoints.

SECONDARY OUTCOMES:
Microbiological profile identified in CSF culture results. | 30 days after study inclusion
  Microbiological characteristics of device-related central nervous system infections, considering the prevalence of microorganisms (multi-resistant or not) at baseline versus the group included after the intervention bundle. The outcome will be measured based on the positive liquor culture and antibiogram.
Risk factors | 30 days after study inclusion
  To compare microbiological characteristics of device-related central nervous system infections, considering the prevalence of microorganisms (multi-resistant or not).
Drug treatment during hospital stay | 30 days after study inclusion
  To compare treatment practices for device-related central nervous system infections at baseline versus the group included after the intervention bundle. The outcome will be measured based on the antibiotic classes used to treat CNS infection, dose and time of use of antibiotics. The treatment data will be collected from the medical prescription during the hospital stay.
Diagnostic accuracy | 30 days after study inclusion
  The difference between the percentages of suspected and confirmed infection cases at baseline will be evaluated, compared to the group included after the intervention bundle.
Cost of hospital admission in dollars, comparing patients with and without infection | 30 days after study inclusion
  Compare costs associated with the duration of infection at baseline versus the group included after the intervention bundle. The outcome will be measured based on the demographic characteristics, Saps3, infection (yes or no), use of antibiotics and time of permanence on ICU.
Death rate | 30 days, 6 months and 1 year after study inclusion
  The outcome will be measured based on the vital status on the hospital discharge, follow-up in 30 days, 6 months and 1 year.
Rankin scale | 30 days, 6 months and 1 year after study inclusion
  Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  The patient is classified as follows:
  * No symptoms at all;
  * No significant disability despite symptoms; able to carry out all usual duties and activities
  * Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  * Moderate disability; requiring some help, but able to walk without assistance
  * Moderately severe disability; unable to walk and attend to bodily needs without assistance
  * Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  * Dead
  Compare rankin scale score before and after the intervention bundle.
Adherence of the study site to the intervention bundle | Monthly
  From the first patient enrollment at participating centers to the last hospital discharge of the recruited sample.

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Veiga, Phd, Principal Investigator — BP - A Beneficência Portuguesa de São Paulo; Renata Oliveira, Principal Investigator — Hospital Geral Clériston Andrade; Cássia Shinotsuka, Principal Investigator — Instituto Estadual do Cérebro Paulo Niemeyer; Thiago Lisboa, Principal Investigator — Hospital de Clinicas de Porto Alegre; Luciana Sanches, Principal Investigator — Hospital do Amor de Barretos; Lívia Medeiros, Principal Investigator — Hospital Pelópidas Silveira; Tássio Lavor, Principal Investigator — Hospital Getúlio Vargas; Débora Pinho, Principal Investigator — Hospital da Restauração; Cristiano Franke, Principal Investigator — Hospital de Pronto Socorro de Porto Alegre; Gabriela Teixeira, Principal Investigator — Hospital Universitário Cajuru; Eliane Silva, Principal Investigator — Hospital Universitário Onofre Lopes; Marcelo Romano, Principal Investigator — Hcor - Associação Beneficente Síria; Wilson Lovato, Principal Investigator — Hospital das Clínicas de Ribeirão Preto; Israel Maia, Principal Investigator — Instituto Baía Sul de Ensino e Pesquisa Irineu May Brodbeck; Priscila Gonçalves, Principal Investigator — Santa Casa de Misericordia de Passos; Flávia Machado, Principal Investigator — Hospital São Paulo; Glécia Rocha, Principal Investigator — Instituto Hospital de Base do Distrito Federal - IGESDF; Roberta Roepek, Principal Investigator — Hospital das Clínicas FMUSP

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Champey J, Mourey C, Francony G, Pavese P, Gay E, Gergele L, Manet R, Velly L, Bruder N, Payen JF. Strategies to reduce external ventricular drain-related infections: a multicenter retrospective study. J Neurosurg. 2018 Jun 22;130(6):2034-2039. doi: 10.3171/2018.1.JNS172486. Print 2019 Jun 1. PMID 29932377
- [Background] Ramanan M, Lipman J, Shorr A, Shankar A. A meta-analysis of ventriculostomy-associated cerebrospinal fluid infections. BMC Infect Dis. 2015 Jan 8;15:3. doi: 10.1186/s12879-014-0712-z. PMID 25567583
- [Background] Jin J, Akau Ola S, Yip CH, Nthumba P, Ameh EA, de Jonge S, Mehes M, Waiqanabete HI, Henry J, Hill A; International Society of Surgery (ISS) and the G4 Alliance International Standards and Guidelines for Quality Safe Surgery and Anesthesia (ISG-QSSA) Group. The Impact of Quality Improvement Interventions in Improving Surgical Infections and Mortality in Low and Middle-Income Countries: A Systematic Review and Meta-Analysis. World J Surg. 2021 Oct;45(10):2993-3006. doi: 10.1007/s00268-021-06208-y. Epub 2021 Jul 3. PMID 34218314
- [Background] Lord AS, Nicholson J, Lewis A. Infection Prevention in the Neurointensive Care Unit: A Systematic Review. Neurocrit Care. 2019 Aug;31(1):196-210. doi: 10.1007/s12028-018-0568-y. PMID 29998427
- [Background] Karvouniaris M, Brotis A, Tsiakos K, Palli E, Koulenti D. Current Perspectives on the Diagnosis and Management of Healthcare-Associated Ventriculitis and Meningitis. Infect Drug Resist. 2022 Feb 28;15:697-721. doi: 10.2147/IDR.S326456. eCollection 2022. PMID 35250284